CLINICAL TRIAL: NCT02847364
Title: Does Chewing Gum Affect the Incidence of Post-operative Ileus in Patients Undergoing Spine Surgery?
Brief Title: Effect of Chewing Gum on Post-operative Ileus (GUMPI)
Acronym: GUMPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Abdel Majid Sheikh Taha, Clinical Instructor of Orthopedic Surgery, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SUR.AMST.01
Record Dates: First submitted 2016-07-15; First posted 2016-07-28 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Ileus
Keywords: chewing gum; prevention
MeSH Terms: conditions — Ileus | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chewing gum group (Experimental): The patients will be asked to chew on a regular chewing gum starting morning of post-operative day 1 until the first bowel movement.
  Interventions: Dietary Supplement: chewing gum
- Control group (No Intervention): These patients will not be offered any food/beverage orally. Patients will be asked not to eat or chew anything till the first bowel movement.

INTERVENTIONS:
Dietary Supplement: chewing gum — The patient will chew one piece (1.45g) of regular chewing gum starting morning of post-operative day 1 for 30 minutes each time, three times per day, till the first bowel movement.
  Arms: Chewing gum group

SUMMARY:
The purpose of this study is to determine whether chewing gum post-operatively decreases the time to first flatus or defecation in patients undergoing spine surgery as a indirect indicator of post-operative ileus.

DETAILED DESCRIPTION:
The patients undergoing spine surgery are at risk of developing post-operative ileus, which will lengthen the hospital stay and cause gastrointestinal distress in patients. Post-operative sham feeding in form of chewing a gum seems to increase the functionality of gastro-intestinal tract earlier in patients who have undergone gastro-intestinal and gynecological surgeries.

This study will recruit patients undergoing spine surgery at the investigators medical center and allocate them randomly into two equal groups. Patients in one group will be asked to chew gum after surgery and the other group will not be offered anything on chew on. Both groups will be kept nothing per os (NPO) otherwise till the first bowel movement. The first post-operative flatus and defecation time will be recorded as primary measures and other main outcomes will include first post-operative meal, length of stay and presence of ileus. The descriptive parameters of the two groups will also be recorded as related to relevant medical history, surgery, and post-operative care, to adjust for its effect on outcome measures.

This study will identify any beneficial effect that chewing gum will have on post-operative ileus development and might be helpful in establishing better post-operative care protocols in patients undergoing spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient 13 years of age or older
* Patients who will undergo spine decompression, laminectomy (cervical, lumbar and/or thoracic), discectomy, foraminotomy, or corpectomy, with or without arthrodesis, with or without instrumentation.

Exclusion Criteria:

* Less than 13 years of age
* Patients who have undergone with abdominal surgery within the last month
* Patients with inability or problems with chewing and/or dysphagia
* Patients who are expected to be kept intubated after surgery
* Patients who are allergic to any chewing gum component

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2023-02 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
first flatus time | post-operative hospital stay till discharge (up to 5 days)
  time of passing the first flatus after surgery; monitored for first flatus for up to 5 days after surgery.
first defecation time | post-operative hospital stay till discharge (up to 5 days)
  time of passing the first defecation after surgery, monitored for first defecation for up to 5 days after surgery.

SECONDARY OUTCOMES:
LOS | hospital stay (average of 5 days)
  the length of hospital stay (throughout their hospital stay, average of 5 days)
Meal time | post-operative hospital stay till discharge (up to 5 days)
  The time of first tolerable meal after surgery; monitored for first tolerable meal for up to 5 days after surgery.
post-operative ileus | post-operative hospital stay till discharge (up to 5 days)
  presence of post-operative ileus; monitored for ileus for up to 5 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Abdel Majid Sheikh Taha, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jennings JK, Doyle JS, Gilbert SR, Conklin MJ, Khoury JG. The Use of Chewing Gum Postoperatively in Pediatric Scoliosis Patients Facilitates an Earlier Return to Normal Bowel Function. Spine Deform. 2015 May;3(3):263-266. doi: 10.1016/j.jspd.2014.12.001. Epub 2015 Apr 23. PMID 27927468
- [Background] Short V, Herbert G, Perry R, Atkinson C, Ness AR, Penfold C, Thomas S, Andersen HK, Lewis SJ. Chewing gum for postoperative recovery of gastrointestinal function. Cochrane Database Syst Rev. 2015 Feb 20;2015(2):CD006506. doi: 10.1002/14651858.CD006506.pub3. PMID 25914904
- [Background] Zhu YP, Wang WJ, Zhang SL, Dai B, Ye DW. Effects of gum chewing on postoperative bowel motility after caesarean section: a meta-analysis of randomised controlled trials. BJOG. 2014 Jun;121(7):787-92. doi: 10.1111/1471-0528.12662. Epub 2014 Mar 14. PMID 24629205
- [Background] Fineberg SJ, Nandyala SV, Kurd MF, Marquez-Lara A, Noureldin M, Sankaranarayanan S, Patel AA, Oglesby M, Singh K. Incidence and risk factors for postoperative ileus following anterior, posterior, and circumferential lumbar fusion. Spine J. 2014 Aug 1;14(8):1680-5. doi: 10.1016/j.spinee.2013.10.015. Epub 2013 Oct 31. PMID 24184650